CLINICAL TRIAL: NCT06175507
Title: Efficacy of Baclofen Vs Naltrexon in Achieving & Maintaining Abstinence in Alcohol Dependence.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ALD-02
Record Dates: First submitted 2023-11-16; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-10

CONDITIONS: Alcohol Liver Disease
MeSH Terms: interventions — Naltrexone; Baclofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naltrexone (Experimental): Naltrexone 50mg orally once daily will give for 12 weeks
  Interventions: Drug: Naltrexon
- Baclofen (Active Comparator): Baclofen 10mg orally thrice daily will give for 12 weeks
  Interventions: Drug: Baclofen

INTERVENTIONS:
Drug: Naltrexon — Naltrexone 50mg orally once daily will give for 12 weeks
  Arms: Naltrexone
Drug: Baclofen — Baclofen 10mg orally thrice daily will give for 12 weeks
  Arms: Baclofen

SUMMARY:
ALD is the most common cause of liver cirrhosis in western world. In patients with ALD persistent alcohol intake is associated with increased mortality while cessation of alcohol consumption improve survival. Baclofen is GABA-B receptor agonist and it is safe in cirrhotic patient for alcohol abstinence i.e. already proven and naltrexone is Delta and k-opioid receptor antagonist and it is safe in cirrhotic for alcohol abstinence i.e, proven in ILBS.

DETAILED DESCRIPTION:
Aim and Objective:

• To compare the efficacy of Naltrexone Vs Baclofen in achieving and maintaining 12-week abstinence in patients with alcohol associated liver cirrhosis with continued alcohol use

Primary objective:

* The comparison in the proportion of patients achieving and maintaining alcohol abstinence between Naltrexone and Baclofen in alcohol associated liver cirrhosis patients with continued alcohol intake at 12 weeks
* Secondary objectives:

  * To evaluate drinking pattern before and after 4 week on Naltrexone without liver related adverse effects compared to baclofen
  * To evaluate proportion of patients maintaining abstinence from alcohol in both the group at 24 weeks
  * To evaluate difference in craving measures between groups at 4, 8,12 and 24 weeks
  * To evaluate difference in alcohol free days between groups at 4, 8,12 and 24 weeks
  * To evaluate proportion of patients developing lapse and relapse in both the group at 4,8,12 and 24 weeks
  * To evaluate the progression of liver disease in both group

Methodology:

* Study population: All patients aged ≥ 18 years and ≤ 65 years admitted in Institute of Liver and Biliary Sciences, New Delhi with alcohol dependence in compensated liver disease and are giving written consent for participation in the study.
* Study design - Single center, Open label, Randomized controlled trial
* Study period - 1.5 years after IEC approval.
* Sample size - We are enrolling 110 patients, with 55 in each arm.
* Intervention -
* Naltrexon group: Naltrexone 50mg orally once daily will give for 12 weeks.
* Baclofen group: Baclofen 10mg orally thrice daily will give for 12 weeks.
* Monitoring and assessment:
* Follow up- weekly in first month and 2nd weekly there after
* LFT (AST, ALT, GGT, Albumin, INR), CBC with MCV, KFT at every visit At every visit
* Review of drinking and assessment of abstinence, lapses and relapses from alcohol
* Overall functioning, quality of life, social relationships
* Difficulties with treatment adherence (pill counts)
* Adverse effects - drug/ withdrawal related
* Psychological support and counselling at every visit by psychiatrist
* Statistical Analysis: The data will be represented as mean±SD. The categorical data will be analysed using Chi-square test. The continuous data will be analysed by student T test, or Mann-Whitney test, whichever is applicable. Besides this, Cox regression will be applied to analyse the variables. For all tests, p≤ 0.05 will be considered statistically significant
* Adverse effects
* Headaches, nausea, dyspepsia, anorexia, anxiety and sedation.
* Stopping rule
* Worsening of liver disease severity to CTP >9
* AST or ALT > 5 times ULN
* Withdrawal of consent
* New onset decompensation
* Worsening of Bilirubin > 5 mg/dl

Expected outcome of the project:

- To achieve abstinence in both the group without affecting the liver.

ELIGIBILITY:
Inclusion Criteria:

1. All consecutive alcohol related compensated cirrhotic patients with continued alcohol consumption despite counselling in last 4 weeks aged between 18 - 65yrs
2. Fulfilling DSM - 5 criteria for alcohol use disorder (Association, 2013)
3. History of recent recidivism / relapse

Exclusion Criteria:

1. Current HE
2. Total Bilirubin > 5 mg/dl
3. Recent bleed
4. Treatment with corticosteroids within the past 60 days
5. Unwilling to participate
6. Dependence on any other substance (except Nicotine)
7. Psychotic disorder requiring treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-12-25 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
The comparison in the proportion of patients achieving and maintaining alcohol abstinence between Naltrexone and Baclofen in alcohol associated liver cirrhosis patients with continued alcohol intake at 12 weeks | 12 weeks

SECONDARY OUTCOMES:
To evaluate abstinence rate by OCDS score in both the group (OCDS- Obsessive compulsive drinking scale 0-40, Higher total score indicate more obsessive thoughts or compulsive behaviour regarding alcohol use) | 4 weeks
To evaluate proportion of patients maintaining abstinence from alcohol in both the group at 24 weeks | 24 weeks
To evaluate difference in craving measures between groups at 4,8,12 and 24 weeks. | 4, 8,12 and 24 weeks
  Craving measures will be assessed based on pre existing structured and validated questionnaires. (Visual analogue scale (VAS) score, score 0-10, 10 suggestive of maximum craving).
To evaluate difference in alcohol free days between groups at 4, 8,12 and 24 weeks | 4, 8,12 and 24 weeks
To evaluate proportion of patients developing lapse and relapse in both the group at 4,8,12 and 24 weeks | 4,8,12 and 24 weeks
To evaluate the progression of liver disease in both group at 24weeks by measuring Child pugh score. | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided